CLINICAL TRIAL: NCT07015086
Title: The Effect of Guided Imagery and Positive Birth Experience Sharing on Fear of Childbirth and Self-Efficacy: A Randomized Controlled Trial
Brief Title: Guided Imagery and Positive Birth Experience Sharing on Fear of Childbirth and Self-Efficacy
Acronym: non
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Sidika Pelit Aksu, Assistant professor in the department of obstetrics, gynecology and diseases nursing, Gazi University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: E-77082166-604.01-1251133; non (Other: non)
Record Dates: First submitted 2025-06-03; First posted 2025-06-11 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-06

CONDITIONS: Childbirth
Keywords: birth; guided imagery; birth fear; positive birth experience; self-efficacy
MeSH Terms: interventions — Imagery, Psychotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): Pregnant women will be invited to sessions by forming groups of 3-10 people. A face-to-face positive birth experience sharing and mental visualization practice will be done once in the 26-28th weeks of pregnancy at the Gazi University Health Research and Application Center Gynecology and Obstetrics Polyclinic. The positive experience sharing will be done by one of the researchers personally and the pregnant women's questions will be answered after the sharing. The mental visualization techniques prepared by Rossman (2015) to facilitate birth will be used for the mental visualization practice. After the training, the mental visualization instructions will be given to the pregnant women as an audio recording in mp3 format. The pregnant women will be asked to mentally visualize once or twice a day for at least 10 weeks. The mental visualization practice takes approximately 20 minutes. The pregnant women will be reminded to do the practice every day via the Whatsapp® application.
  Interventions: Behavioral: Guided Imagery and Positive Birth Experience Sharing
- control group (No Intervention): No intervention will be applied to the control group. Post-test and follow-up tests will be applied at the same times and with the same scales as the intervention group. Finally, the method of birth will be questioned.

INTERVENTIONS:
Behavioral: Guided Imagery and Positive Birth Experience Sharing — The positive experience will be shared by one of the researchers and the pregnant women's questions will be answered after the sharing. The mental imagery techniques prepared by Rossman (2015) to facilitate birth will be used for the mental imagery application. After the training, the mental imagery instructions will be given to the pregnant women as an audio recording in mp3 format. The pregnant women will be asked to do the mental imagery once or twice a day for at least 8 weeks. The mental imagery application takes approximately 20 minutes. The pregnant women will be reminded to do the application every day via the Whatsapp® application. The pregnant women will be asked to mark whether they do the application every day or not on the weekly follow-up chart.
  Arms: experimental group

SUMMARY:
Abstract This study will be conducted to determine the effect of sharing positive birth experiences and mental imagery on birth self-efficacy and fear of childbirth. The study is a single-center, parallel-group, stratified block (in terms of fear of childbirth level) randomized controlled experimental study. The study sample will consist of a total of 84 participants, with 42 in the intervention group and 42 in the control group. The study is planned to be conducted between July 1, 2025, and July 1, 2026. Inclusion criteria for the study are: WİJMA A scale score average below 85, age over 18, being primiparous, being in the 20th to 26th week of pregnancy, having no complications in the mother or fetus during pregnancy (gestational diabetes, hypertension, preeclampsia, intrauterine growth restriction, congenital anomalies, etc.), having no communication problems (mental, auditory, visual, language, etc.), and volunteering to participate in the study. The study data will be collected using a personal information form, the Wijma Childbirth Expectancy/Experience Scale Version A (W-DEQ A), and the Childbirth Self-Efficacy Scale-Short Form (CBSEI-C32). Women will be invited to participate in online training sessions in groups of 3-10 people. Positive birth stories will be shared with the women, and visualization exercises will be demonstrated. Following the training sessions, the follow-up phase of the study will begin, and women will be provided with an audio recording of the visualization guidelines in MP3 format. Women will be asked to perform visualization exercises at least once or twice daily for a minimum of eight weeks. No intervention will be applied to the control group.

DETAILED DESCRIPTION:
Problem Definition Cesarean delivery has significant benefits in high-risk pregnancies, but unnecessary and excessive use of cesarean section has negative consequences on the physical, emotional, and mental health of both mothers and babies. It also places an increasing financial burden on the healthcare system . The increase in the rate of planned cesarean sections before birth cannot be explained by clinical risk factors. This situation can be explained by mothers' preference for planned cesarean sections.

Women's preferences for cesarean sections before birth are influenced by social and cultural factors as well as psychological factors. The most commonly reported psychological factors associated with birth preferences are birth self-efficacy and fear of childbirth. Birth self-efficacy is defined as a person's belief that they can cope with the act of childbirth and the vaginal birth process. Carlson et al. reported that nulliparous women with low self-efficacy in the third trimester of pregnancy experienced higher levels of fear of childbirth compared to women with high self-efficacy. In another study, Lowe found that nulliparous women with lower childbirth self-efficacy were more likely to plan for a cesarean delivery compared to those with higher childbirth self-efficacy. In a study by Schwartz and colleagues, it was determined that self-efficacy is significantly associated with birth preference, independent of parity, and that the intention to have a cesarean delivery increases as self-efficacy decreases. Reducing fear of vaginal birth, thereby increasing positive perceptions of vaginal birth, is important in reducing cesarean preferences.

Having a positive birth experience with vaginal birth or hearing about someone else's positive birth experience can be effective. The sharing of birth stories has increased with the development of new technologies, and women can more easily access others' birth stories through multimedia platforms. Carlsson et al. reported that 97% of nulliparous women had heard birth stories from their mothers and friends. Amyx et al. noted that birth stories are the third most important source of information for nulliparous women, after healthcare professionals and prenatal classes. In a qualitative study of nulliparous women, birth stories were identified as the most useful source of information by 71% of women. Regardless of the type of birth, birth stories have a strong effect on self-efficacy and fear. Therefore, listening to positive birth stories may reduce birth fear in pregnant women.

In recent years, relaxation techniques aimed at reducing fear of childbirth have been increasingly used. One such relaxation technique, mental imagery, is a method for treating stress and anxiety by replacing distressing memories with positive mental images. This involves instructional guidance that triggers sensory experiences, behavioral, and physiological responses. Boryri et al. (2019) found that visualization was effective in reducing fear of childbirth in pregnant women to prevent planned and unnecessary cesarean sections. This study will be conducted to determine the effect of positive birth experience sharing and visualization on birth self-efficacy and fear of childbirth.

ELIGIBILITY:
Inclusion Criteria:

* The WIJMA A scale score average should be below 85, be over 18 years of age, be primiparous, be in the 20-26th week of pregnancy, not have any complications in the mother or fetus during pregnancy (gestational diabetes, hypertension, preeclampsia, intrauterine growth retardation, congenital anomaly, etc.), not have any communication problems (mental, auditory, visual, language, etc.), and be willing to participate in the study.

Exclusion Criteria:

* Failure to perform post-tests,
* Participant's wish to withdraw from the study at any stage of the study,
* Pregnancy turning into a risky pregnancy,
* Birth occurring before the 37th week of pregnancy,
* Not performing the visualization exercise for at least three consecutive days.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2025-08-25 (Estimated); Primary Completion 2026-05-25 (Estimated); Study Completion 2026-12-12 (Estimated)

PRIMARY OUTCOMES:
Difference of scores of the Wijma Childbirth Expectation/Experience Scale Version A | 8 weeks
  There is a difference between the intervention and control groups in terms of the mean post-test scores of the Wijma Childbirth Expectation/Experience Scale Version A. The minimum score that can be obtained from the scale is 0, and the maximum score is 165. High scores indicate that women have a high fear of childbirth. W-DEQ A score ≤37 indicates mild, 38-65 indicates moderate, 66-84 indicates severe, and ≥85 indicates clinical level fear.
Difference of scores of the Labor Self-Efficacy Scale-Short Form. | 8 weeks
  There is a difference between the intervention and control groups in terms of the mean post-test scores of the Labor Self-Efficacy Scale-Short Form.The scale has two sub-dimensions: outcome and adequacy expectations. Each sub-dimension of the scale consists of 16 questions. The lowest score that can be obtained from the scale sub-dimensions is 16, and the highest score is 160. A high score obtained from the sub-dimensions indicates that pregnant women have high adequacy and outcome expectations regarding birth. Responses on the Likert-type scale are scored from 1 to 10. The lowest total score that can be obtained from the scale is 32, and the highest score is 320. High scores obtained from the scale indicate that pregnant women have high levels of self-efficacy in labor.

CONTACTS AND LOCATIONS:
Locations (1):
- Nursing Faculty of Gazi University, Ankara, Turkey, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No